CLINICAL TRIAL: NCT00172107
Title: A Double Blind, Placebo Controlled, Parallel-Group Study to Assess the Safety and Efficacy of 3 Doses of ALX1-11 (50, 75, and 100µg) in the Treatment of Postmenopausal Osteoporosis
Brief Title: A Study to Assess the Safety and Efficacy of 3 Doses of ALX1-11 (50, 75, and 100µg) in the Treatment of Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: CL1-11-821
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Osteoporosis
Keywords: Post-menopausal; Osteoporosis; Parathyroid Hormone; PTH; ALX1-11
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo drug injectable subcutaneously
  Interventions: Drug: placebo
- 2 (Experimental): 50 mcg PTH(1-84)
  Interventions: Drug: ALX1-11 50 mcg
- 3 (Experimental): 75mcg PTH(1-84)
  Interventions: Drug: ALX1-11 75mcg
- 4 (Experimental): 100 mcg PTH(1-84)
  Interventions: Drug: ALX1-11

INTERVENTIONS:
Drug: ALX1-11 50 mcg — PTH(1-84) 50 mcg for subcutaneous injection into thigh or abdomen
  Other Names: PREOS
  Arms: 2
Drug: placebo — placebo powder for subcutaneous injection
  Arms: 1
Drug: ALX1-11 75mcg — PTH(1-84)75 mcg for subcutaneous injection
  Other Names: PREOS
  Arms: 3
Drug: ALX1-11 — PTH (1-84) 100mcg for subcutaneous injection into thigh or abdomen
  Other Names: PREOS
  Arms: 4

SUMMARY:
A double-blind, placebo-controlled, parallel-group study to assess the safety and efficacy of 3 doses of ALX1-11 (recombinant human parathyroid hormone [rhPTH(1-84)])(50, 75 and 100 µg) in the treatment of postmenopausal osteoporosis. The primary objective of this study is to compare the efficacy of ALX1-11 (50, 75 and 100 µg) with that of placebo in terms of increasing vertebral bone mineral density, when given daily by subcutaneous injection for 12 months in postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
Human clinical experience with a synthetic human parathyroid hormone fragment (rhPTH 1-34) and animal studies with ALX1-11 demonstrate consistent increases in bone mineral density. Furthermore, the newly formed bone is normal in structure and composition. Therefore, ALX1-11 (recombinant human parathyroid hormone [rhPTH 1-84]) has the potential to stimulate new bone formation in osteoporotic patients thereby increasing trabecular bone density and preventing fractures. The clinical profile for ALX1-11 can be expected to be unique, since none of the approved therapies for osteoporosis are able to form the quantities of new bone that ALX1-11 is potentially capable of. Patients with bone density below the "fracture threshold" (osteopenia), as well as those with established vertebral fractures (osteoporosis), would be expected to benefit from treatment.

Animal toxicology studies have been completed and there were no results to indicate any restrictions in the clinical usage of the drug. Preliminary human clinical experience with ALX1-11 in healthy, postmenopausal females has demonstrated no apparent risk of frank hypercalcemia* at single administrations up to 5.0 µg/kg or daily administrations for 7 days up to 2.0 µg/kg/day.

Based on these studies, the anticipated therapeutic range of ALX1-11 is 50-100 µg per day (approx. 1.0 - 1.5 µg/kg/day). Therefore, the dose range to be tested in this study will include an anticipated minimally effective dose, interim dose and maximally tolerable dose (50, 75 and 100 µg). The efficacy of 3 doses of ALX1-11 will be assessed in terms of bone mineral density and biochemical markers of bone turnover in postmenopausal women.

The primary objective of this study is to determine the dose-response relationship of ALX1-11 in terms of bone mineral density. The efficacy of the 3 doses of ALX1-11 relative to placebo will be determined by measurement of bone mineral density (by DXA) at baseline and at 3, 6 and 12 months.

Patients will administer a daily subcutaneous injection of 0.5 mL of either 50, 75 or 100 µg of ALX1-11 or placebo every morning for 12 months.

Women will be advised to use the provided calcium supplements (500mg elemental calcium) to maintain a total daily intake of 1000-1500 mg/day and vitamin D supplements will also be provided (400 IU/day). A dietary questionnaire will be done at visit screen, 6 and 15.

If a patient's total serum calcium measurement, during the treatment phase, demonstrates frank hypercalcemia OR if her pre-dose calcium levels are more than 0.5 mg/dL or 0.125 mmol/L above the upper limit of normal (2.78 mmol/L or 11.1 mg/dL), then the patient's serum calcium level must be repeated.

If upon re-test a patient continues to demonstrate frank hypercalcemia OR if her basal pre-dose calcium levels continues to be elevated above the upper limit of normal, then the patient will be withdrawn from the study.

*Frank Hypercalcemia: defined as total serum calcium levels above 11.1 mg/dL or 2.78 mmol/L

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women aged 50-75 years at Visit 1 (at least 5 years post cessation of menses, or FSH>20 IU/L, serum estradiol <110 pmol/L)
* Vertebral bone mineral density at least 2.5 S.D. below the mean of young normals. Patients must have at least 2 measurable contiguous vertebral bodies in the lumbar region, L1-L4.
* Ability to self administer injections
* Ability and willingness to give informed consent

Exclusion Criteria:

* Evidence of 5 or more vertebral fractures
* Evidence of 2 or more vertebral fractures in the region L1-L4
* Presence of significant cardiac disease as determined by history, physical examination and laboratory screens e.g. cardiac dysrhythmias.
* Presence of significant hepatic, renal, pulmonary, gastrointestinal, hematological, endocrine, immunologic, neurological or psychiatric disease as determined by history, physical examination and laboratory screens. Specifically excluded are diseases known to contribute to osteoporosis: hyperparathyroidism, hyperthyroidism, glucocorticoid excess, hyper or hypocalcemia, Paget's disease, osteogenesis imperfecta, osteomalacia and severe scoliosis.
* Evidence of lumbar fusions, osteophytes or excessive degenerative disease which precludes reasonable DXA measurement.
* History or presence of cancer within the previous 5 years except for superficial basal cell and squamous cell carcinomas of the skin.
* Treatment with any of the following therapies:

  * Any form of Estrogen within previous 6 months
  * Prior use of Etidronate for more that 2 treatment cycles (2weeks/cycle) and/or any use within prior 6 months
  * Any other bisphosphonate
  * Parathyroid Hormone use within 6 months
  * Fluoride (>10 mg/day) within 12 months
  * Any form of Calcitonin within previous 4 months
  * Thyroid hormone within previous 4 months unless TSH levels found to remain within normal range
  * Other therapies known to influence bone metabolism* within previous 4 months
  * Any investigational compound within previous 3 months
  * Abnormal serum Ca++ level: patients having two (2) consecutive serum calcium above 2.66 mmol/L (10.6 mg/dl) will be excluded.
  * History of positive test for Hepatitis B or C, or urine drug screen.
  * History of alcohol or drug abuse: an excess of alcohol is defined as more than 4 or any combination of more than four (4) of the following per day: 120 mL wine, 360 mL beer or wine cooler or 30 mL whiskey.
  * Weight more than 25% above ideal body weight, (minimum 45 kg) as listed in the Metropolitan Life Insurance Tables (Appendix 3)
  * Deemed unsuitable, in the opinion of the investigator, for any other reason.

(*Chronic or continued use of medication that may affect bone calcium metabolism, e.g. thiazide diuretics, oral or injectable steroids, antimitotics (methotrexate), heparin, anticonvulsants and supplements of Vitamin D in excess of 1,000 IU per day and Vitamin A in excess of 10,000 IU per day)

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 1995-05-18 (Actual); Primary Completion 1997-03-24 (Actual); Study Completion 1997-03-24 (Actual)

PRIMARY OUTCOMES:
Efficacy was assessed as percent change from baseline in BMD, BMC, and BMA at the lumbar spine, total hip, femoral neck and whole body (excluding the head) using DXA. | 12 months of treatment

SECONDARY OUTCOMES:
Secondary efficacy evaluations were also performed at Month 3, 6, and 12: Percent change from baseline in lumbar spine BMC and BMA; Percent change from baseline in total hip and femoral neck BMD, BMC and BMA | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (19):
- United States (15):
  - Pivotal Research, Peoria, Arizona
  - Loma Linda Osteoporosis Research Clinic, Loma Linda, California
  - Steven Harris, Mill Valley, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Paul Miller, Lakewood, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - Radiant Research, Stuart, Stuart, Florida
  - Maine Center for Osteoporosis Research and Education of St. Joseph's Hospital, Bangor, Maine
  - 'Bethesda Health Research Center, Bethesda, Maryland
  - Helen Hayes Hospital, West Haverstraw, New York
  - Oregon Osteoporosis Center, Portland, Oregon
  - Simona Scumpia, Austin, Texas
  - Radiant Research, Dallas, Dallas, Texas
  - 'Diabetes & Glandular Disease Research Associates, P.A., San Antonio, Texas
  - Northwest Lipid Research Center, Seattle, Washington
- Canada (4):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - Osteoporosis Research Center, Vancouver, British Columbia
  - Capital Health Centre, Halifax, Nova Scotia
  - St. Joseph's Health Center, London, Ontario